CLINICAL TRIAL: NCT00786786
Title: Perceived Barriers to Exercise in Individuals Living With Spinal Cord Injury.
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Kimberly Anderson, Assistant Adjunct Professor, University of California, Irvine
Other Study IDs: 2008-6465
Record Dates: First submitted 2008-11-04; First posted 2008-11-06 (Estimated); Last update posted 2010-11-04 (Estimated); Status verified 2010-11

CONDITIONS: Spinal Cord Injury
Keywords: Any person with a spinal cord injury; at least 18 years of age
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Spinal Cord Injury

SUMMARY:
Purpose: This project is designed to identify what the key barriers to participating in exercise are for the general population of people living with spinal cord injury (SCI) in the United States (US).

DETAILED DESCRIPTION:
Purpose: This project is designed to identify what the key barriers to participating in exercise are for the general population of people living with spinal cord injury (SCI) in the United States (US).

Background: A previous study of 681 people living with SCI demonstrated that the majority of participants thought that exercise was important (97%), but that only 57% actually had access to exercise (K.D. Anderson. 2004. Targeting recovery: Priorities of the spinal cord injured population. J. Neurotrauma. 21:1371-1383). The next step in continuing that research is to determine in more detail what the perceived barriers to exercise are so that they can be addressed in multiple settings (research design of exercise protocols, community access and awareness, clinical effectiveness, etc.).

Methods: Internet-based survey of people with spinal cord injuries (SCI). Expected Results: It is expected that the perceived barriers will fall under 3 main categories (internal, resources, and structural). However, there may be other barriers we are unaware of, for example, societal or cultural factors or other factors completely unforeseen.

Relevance to Rehabilitation: The findings of this project will provide valuable information needed to design strategies aimed at improving participation in exercise by people living with SCI. SCI results in several secondary health conditions over time, which can likely be positively impacted by exercise.

ELIGIBILITY:
Inclusion Criteria:

* Any person with a spinal cord injury who is at least 18 years of age, lives in the United States of America, and can read English.

Exclusion Criteria:

* People who cannot read English will not be included because the website will be hosted in English and the survey software (phpQuestionnaire 2.2 by Chumpsoft, Inc.) default language is English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any person with a spinal cord injury who is at least 18 years of age, lives in the United States of America, and can read English.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2008-08; Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Anderson, Ph.D., Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States